CLINICAL TRIAL: NCT04994496
Title: Evaluation of a Web-based Self-help Intervention Based on Principles of Positive Psychology Promoting Mental Health in Adolescents
Brief Title: Web-based Self-help Intervention Promoting Mental Health in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Prof. Otto Beisheim Foundation (Other)
Responsible Party: Principal Investigator, Ellen Greimel, Postdoctoral Researcher, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20115
Record Dates: First submitted 2021-07-30; First posted 2021-08-06 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Mental Health; Positive Thinking; Stress; Depressive Symptoms
Keywords: Mental Health; Adolescence; Youth; Prevention; Positive Psychology; Self-help; Web-based Intervention
MeSH Terms: conditions — Psychological Well-Being; Depression

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups in parallel for the duration of the study
Who Masked: Participant
Masking Description: Participants are not aware of the assigned intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based intervention group (Experimental): Two-week web-based intervention group
  Interventions: Behavioral: Two-week web-based self-help intervention based on principles of positive psychology
- Web-based control group (Sham Comparator): Two-week web-based sham comparator
  Interventions: Behavioral: Two-week web-based text messages containing fun facts

INTERVENTIONS:
Behavioral: Two-week web-based self-help intervention based on principles of positive psychology — The web-based self-help intervention consists of 14 exercises based on the following positive psychology domains: personal strengths, pleasure, gratitude, engagement (flow, mindfulness) and positive relationships.
  The (partly interactive) exercises are created to be implemented by the participants themselves without support of a therapist.
  Before starting the intervention, the participants are told that they will receive a daily email with an instruction for a short exercise over the period of two weeks. The participants are instructed to complete the exercises every day and are told that they will be asked to evaluate these exercises at the next appointment (post-test, week 2)
  Arms: Web-based intervention group
Behavioral: Two-week web-based text messages containing fun facts — The web-based sham intervention consists of 14 text messages containing random interesting facts ("fun facts").
  Before starting the sham intervention, the participants are told that they will receive a daily email with a text message to read every over the period of two weeks. The participants are instructed to read these text messages every day and are told that they will be asked to evaluate these exercises at the next appointment (post-test, week 2)
  Arms: Web-based control group

SUMMARY:
This study aims to evaluate the feasibility and effectiveness of a web-based self-help intervention promoting mental health in adolescents. We will examine whether this intervention improves positive affect, reduces stress and alleviates negative affect and depressive symptoms in adolescents aged 12 to 18 years. We will also investigate the rates of adherence among the adolescents who use this web-based intervention and the acceptability of the intervention with adolescents.

DETAILED DESCRIPTION:
The prevalence of mental health problems including depression rises during adolescence. Nevertheless, young people often have little knowledge about mental health problems and conditions, such as depression, and how they can be prevented. Besides limited knowledge, concerns about social stigma, confidentiality and limited access to mental health services are some of the main barriers to seek help. Therefore, highly acceptable and easily accessible services promoting mental health, such as knowledge about mental health conditions and effective self-help strategies to prevent them, are urgently needed for adolescents.

We developed a website, which provides evidence-based information about depressive disorders in youth (e.g., identification, etiology, treatment, and prevention of depression) and will be launched in autumn 2021. Furthermore, the website provides information about self-help strategies (e.g., reducing stress, doing exercise, undertaking positive activities), which are meant to serve as an addition to professional treatments of depression or to promote mental health in adolescents. Target groups of the website are adolescents aged 12 to 18 years seeking help for depression, as well as healthy adolescents seeking information about mental health promotion or prevention of depression.

To increase the acceptability of the website and the engagement of young people, the website will integrate continuously updating content consisting of short exercises based on principles of positive psychology. This web-based self-help intervention is thought to provide a mode of delivery (the combination: "online" & "positive psychology"), which is acceptable and engaging to youth, and might effectively promote mental health in adolescents.

Since the website targets two different groups, we will evaluate the web-based self-help intervention accordingly:

Target group 1: Adolescents with a major depressive disorder (acute or remitted) Target group 2: Healthy Adolescents (no mental health condition)

The current study will focus on target group 2. A study focusing on target group 1 can be found in a separately registered clinical trial on clinicaltrials.gov.

The primary aim of the study is to evaluate the feasibility and effectiveness of this web-based self-help intervention to improve positive affect, reduce stress, alleviate negative affect and depressive symptoms in adolescents.

Participating young people will be randomized to either the web-based intervention group or a web-based control group (i.e. sham intervention / comparator). All participants will be evaluated at pre-, post-intervention, and at a two-week follow-up.

Hypothesis: Participants in the web-based intervention group will report a significant decrease of negative affect, depressive symptoms and perceived stress compared to participants in the web-based control group. Participants in the web-based intervention group will report a significant increase of positive affect compared to participants in the web-based control group

ELIGIBILITY:
Inclusion Criteria:

* Intelligence quotient (IQ) of ≥ 80

Exclusion Criteria:

* Current diagnosis of a mental disorder
* Remitted depressive disorder
* Insufficient knowledge of German

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Affect Schedule for Children-Short Form (PANAS-C-SF) | Pre-test (week 0), post-test (week 2), follow-up (week 4)
  The PANAS is a self-report inventory to assess positive and negative affect (10 items for PA and 10 items for NA), rated on a 5-point response scale, with higher scores indicating more positive affect or negative affect. Participants will complete the PANAS at pre-, post-test and follow-up to determine change in negative and positive affect
Beck Depression Inventory - Second Edition (BDI-II) | Pre-test (week 0), post-test (week 2), follow-up (week 4)
  The BDI-II is a self-report inventory to assess the severity of depressive symptoms, rated on a 4-point response scale, with higher scores indicating more severe depressive symptoms. Participants will complete the BDI-II at pre-, post-test and follow-up to determine change in depressive symptoms
Perceived Stress Scale (PSS-10) | Pre-test (week 0), post-test (week 2), follow-up (week 4)
  The PSS-10 is a self-report inventory to assess perceived stress, rated on a 5-point response scale, with higher scores indicating more perceived stress. Participants will complete the PSS-10 at pre-, post-test and follow-up to determine change in perceived stress

SECONDARY OUTCOMES:
Adherence | Post-test (week 2)
  A self-report inventory, designed by the investigators, to measure the rate of adherence to the intervention
Acceptance | Post-test (week 2)
  A self-report inventory, designed by the investigators, to measure the acceptability / appeal of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Schulte-Körne, Professor, Study Director — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University Hospital Munich
Locations (1):
- Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University Hospital Munich, Munich, Germany, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Data in our study contains sensitive patient information, such as sociodemographic information and comorbidities. Since patients could possibly be identified by making our raw data publicly available, ethical principles of protecting patient confidentiality would be breached. Aggregated group data can be made available upon request

REFERENCES:
- [Derived] Kaubisch S, Kloek M, Primbs R, Iglhaut L, Piechaczek CE, Keim PM, Feldmann L, Schulte-Korne G, Greimel E. A web-based approach to adolescent mental health: Randomized controlled trial of a brief Positive Psychology intervention. Internet Interv. 2025 Sep 12;42:100872. doi: 10.1016/j.invent.2025.100872. eCollection 2025 Dec. PMID 41141290